CLINICAL TRIAL: NCT04265755
Title: Biomarker and Genetic Predictors of Erenumab Treatment Response, a Phase 4 Investigational Open-label Study (INTERROGATE)
Brief Title: Biomarker and Genetic Predictors of Erenumab Treatment Response
Acronym: INTERROGATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190006; 2019-002331-28 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: Migraine
Keywords: Episodic and Chronic Migraine; Link between clinical response and biomarker; Phase 4
MeSH Terms: conditions — Migraine Disorders; Recurrence | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Erenumab packed in a SureClick® Autoinjector Pen (AI)
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Erenumab 70 mg or 140 mg packed in a SureClick® Autoinjector Pen (AI).
  Other Names: AIMOVIG

SUMMARY:
To explore the relationship between clinical response to erenumab and genetic biomarkers

DETAILED DESCRIPTION:
This is a phase 4 open-label study aiming to explore the relationship between clinical response to erenumab and genetic biomarkers.

Subjects with episodic or chronic migraine will be treated with Erenumab 70mg or 140mg for a 4-week baseline/screening period, followed by a 24-week treatment period.

Subjects will collect migraine-related parameters daily using an eDiary and blood samples will be collected for biomarker research. All analysis will be descriptive in nature.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age greater than or equal to 18 years upon entry into screening
* History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self report
* Greater than or equal to 4 headache days that meet criteria as migraine days per month on average across the 3 months before screening After baseline period
* Must have demonstrated greater than or equal to 75% compliance in eDiary usage during baseline period

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

Disease Related

* Greater than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine headache
* Inability to differentiate between migraine from other headaches. Other Medical Conditions
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behaviour
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Prior/Concomitant Therapy

* Previously received erenumab (Aimovig®)
* Received an anti-CGRP monoclonal antibody within 3 months prior to the start of the baseline period
* Initiation, discontinuation, or change of dosing of migraine prophylactic medications within 2 months prior to the start of the baseline period, during the baseline period or planned during the study.

Prior/Concurrent Clinical Study Experience

• Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives since ending treatment on another investigational device or drug study (ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions

* Female subjects of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 16 weeks after the last dose of investigational product
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 16 weeks after the last dose of investigational product
* Evidence of current pregnancy or breastfeeding per subject self-report or medical records
* Subject has known sensitivity to any of the products or components to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1406 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- Glostrup Hospital, Glostrup Municipality, Denmark
- Thjonustumidstod Rannsoknaverkefna, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1406 participants were enrolled in Denmark and Iceland between October 2020 and January 2023.
  As pre-specified, the primary objective of the study was to assess the relationship between migraine polygenic risk score (mPRS) and the reduction in mean monthly migraine days (MMD) after using erenumab, regardless of erenumab dose received.
Pre-assignment Details: The study consisted of the following:
  * A Screening Period of up to 3 weeks.
  * A Baseline Period of 4 - 5 weeks to collect data on migraine headaches and acute headache medication use.
  * A 24-week, Open-label Treatment Period.
Groups:
- Erenumab 70 mg/140 mg: Participants were enrolled into the Open-label Treatment Period and received erenumab 70 mg or 140 mg administered subcutaneously (SC) once every 4 weeks (Q4W) at the discretion of the investigator. Per protocol, dose switching between erenumab 70 mg and 140 mg was permitted at Week 12. However, participants could switch dose before or after Week 12 if needed based on investigator discretion.
  Dose comparison was not pre-specified.
Period: Overall Study
Arm/Group | Erenumab 70 mg/140 mg
Started | 1406
Dose Switch From Baseline Dose | 504
Completed (Completed study) | 1353
Not Completed | 53
Not completed — Withdrawal by Subject | 39
Not completed — Decision by sponsor | 2
Not completed — Lost to Follow-up | 11
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): consisted of all participants who were enrolled in the study.
Groups:
- Erenumab 70 mg/140 mg: Participants were enrolled into the Open-label Treatment Period and received erenumab 70 mg or 140 mg administered SC Q4W at the discretion of the investigator. Per protocol, dose switching between erenumab 70 mg and 140 mg was permitted at Week 12. However, participants could switch dose before or after Week 12 if needed based on investigator discretion.
  Dose comparison was not pre-specified.
Arm/Group | Erenumab 70 mg/140 mg
Number analyzed (Participants) | 1406
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1228
  Male | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 1384
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 17
  Black or African American | 2
  Multiple | 9
  Native Hawaiian or Other Pacific Islander | 0
  White | 1353
  Other | 23
MMDs During the Baseline Period [Mean (Standard Deviation); unit: days / month] — A migraine day was defined as a calendar day (00:00 to 23:59) in which the participant reported any migraine headache or took any triptan-based acute migraine-specific medication. MMDs were calculated as the number of migraine days in the 4 - 5 week Baseline Period.
  days / month | 12.82 (5.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least a 50% Reduction From Baseline in Mean MMDs Over Months 4, 5, and 6 in Relation to mPRS
Description: A migraine day was defined as a calendar day (00:00 to 23:59) in which the participant reports any migraine headache or takes any triptan-based acute migraine-specific medication.
  At least a 50% reduction from Baseline in MMDs was determined if: (average number of migraine days per month during the last 3 months [months 4, 5, and 6] of the 24-week Open-label Treatment Period minus number of migraine days during the 4-week Baseline Period) / number of migraine days during the 4-week Baseline Period * 100, was less than or equal to -50%.
Time Frame: 4-week Baseline Period and the last 3 months (Months 4, 5, and 6) of the 24-week Open-label Treatment Period
Population: Efficacy Analysis Set: consisted of a subset of participants in FAS who received at least 1 dose of investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erenumab 70 mg/140 mg
Number analyzed (Participants) | 1368
percentage of participants | 54.9 [52.22 to 57.56]
Statistical Analysis 1: Comparison: Erenumab 70 mg/140 mg; Odds of achieving at least 50% reduction from Baseline in mean MMD over months 4, 5, and 6 in relation to mPRS; Test type: Other — Adjusted analysis utilizes a logistic regression model which includes age, sex, dose switch, Baseline value of interest, and mPRS as covariates and presents the mPRS estimates; p = 0.86, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.90 to 1.13] — Based on a 1 standard deviation increase in mPRS

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Erenumab 70 mg: Participants who were initially enrolled into the Open-label Treatment Period and received erenumab 70 mg administered SC Q4W at the discretion of the investigator.
- Erenumab 70 mg Switch to 140 mg: Participants who initially received erenumab 70 mg administered SC Q4W and were dose switched to erenumab 140 mg per investigation's discretion.
- Erenumab 140 mg Switch to 70 mg: Participants who initially received erenumab 140 mg administered SC Q4W and were dose switched to erenumab 70 mg per investigation's discretion.
- Erenumab 140 mg: Participants who were initially enrolled into the Open-label Treatment Period and received erenumab 140 mg administered SC Q4W at the discretion of the investigator.
Arm/Group | Erenumab 70 mg | Erenumab 70 mg Switch to 140 mg | Erenumab 140 mg Switch to 70 mg | Erenumab 140 mg
All-Cause Mortality (participants affected / at risk) | 1/214 | 0/497 | 0/7 | 0/688
Serious Adverse Events (participants affected / at risk) | 8/214 | 8/497 | 1/7 | 14/688
Other Adverse Events (participants affected / at risk) | 172/214 | 391/497 | 7/7 | 417/688
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab 70 mg (N=214) | Erenumab 70 mg Switch to 140 mg (N=497) | Erenumab 140 mg Switch to 70 mg (N=7) | Erenumab 140 mg (N=688)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Psychogenic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab 70 mg (N=214) | Erenumab 70 mg Switch to 140 mg (N=497) | Erenumab 140 mg Switch to 70 mg (N=7) | Erenumab 140 mg (N=688)
Constipation (Gastrointestinal disorders) | 92 | 193 | 5 | 280
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 2 | 1 | 7
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Fatigue (General disorders) | 15 | 37 | 0 | 47
Influenza like illness (General disorders) | 12 | 16 | 0 | 14
Injection site bruising (General disorders) | 9 | 34 | 0 | 0
Injection site erythema (General disorders) | 20 | 36 | 0 | 1
Injection site pruritus (General disorders) | 1 | 7 | 1 | 2
Pyrexia (General disorders) | 4 | 6 | 1 | 5
Immunisation reaction (Immune system disorders) | 17 | 35 | 0 | 1
COVID-19 (Infections and infestations) | 49 | 103 | 1 | 57
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 10 | 35 | 0 | 15
Upper respiratory tract infection (Infections and infestations) | 21 | 76 | 0 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | 0 | 3
Dizziness (Nervous system disorders) | 12 | 18 | 0 | 12
Migraine (Nervous system disorders) | 6 | 8 | 1 | 14
Psychogenic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 15 | 14 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 37 | 71 | 1 | 72
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 9 | 3 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04265755/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04265755/SAP_001.pdf